CLINICAL TRIAL: NCT00398008
Title: HIV Risk Reduction and Drug Abuse Treatment in Iran
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never able to start in IRAN
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0207018835; R01DA014718-02S1 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2013-07

CONDITIONS: Opiate Dependence; HIV Infections
Keywords: Buprenorphine; Naltrexone; HIV risk reduction behavior; Counseling; HIV Seronegativity
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections | interventions — Buprenorphine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): DC-HIV plus buprenorphine maintenance.
  Interventions: Drug: Buprenorphine/Subutex; Behavioral: Drug counseling
- 2 (Experimental): DC-HIV plus naltrexone maintenance
  Interventions: Drug: Naltrexone; Behavioral: Drug counseling

INTERVENTIONS:
Drug: Buprenorphine/Subutex — Opioid agonist medication to treat opiate dependence
  Other Names: Subutex
  Arms: 1
Drug: Naltrexone — Opioid antagonist medication to treat opiate dependence
  Arms: 2
Behavioral: Drug counseling — DC-HIV: Drug Counseling that provides education about HIV, drug abuse and dependence; encourages medication adherence; uses motivational enhancement techniques; encourages life style changes; and teaches cognitive and behavioral coping skills to prevent relapse

SUMMARY:
A randomized, double blind clinical trial comparing buprenorphine and naltrexone maintenance treatment when combined with drug abuse and HIV risk reduction counseling (DC-HIV) for heroin and opium addicts in Iran.

DETAILED DESCRIPTION:
This randomized double blind clinical trial compares the efficacy of buprenorphine maintenance treatment (BMT) and naltrexone maintenance treatment (NMT) for recently detoxified opioid dependent patients (N=130; 65 heroin dependent, 65 opium dependent-Specific Aim 1). Manual-guided, HIV risk reduction and drug counseling (DC-HIV) is provided to all patients as the platform psychotherapy. Maintenance treatment is provided for 12 weeks to all patients; patients may also continue to receive maintenance treatment for an additional 12 weeks following the initial treatment period. Primary outcome measures, assessed by twice weekly urine toxicology testing and self-report during the first 12 weeks and monthly during the 12-week extension, include resumption of heroin use, 1 and 3 weeks continuous relapse and reductions in HIV risk behaviors. The project will also evaluate the characteristics of treatment-seeking opioid addicts in Iran (including specific risk behaviors and patterns of HIV risk behaviors; prevalence of psychiatric and other medical comorbidity; and patterns of social, family, vocational, and criminal activity and service needs-Specific Aim 2). This data will be used to revise the DC-HIV manual to address the specific circumstances and risk behaviors of opioid addicts in Iran and to provide data regarding any differential response of opium compared to heroin addicts to BMT or NMT. Finally, the project will also provide clinical training for health professionals and training and mentoring in drug abuse treatment and HIV prevention research to clinical researchers who will continue development, implementation, evaluation and dissemination of HIV prevention and drug abuse treatment approaches in Iran after the project ends (Specific Aim 3). The Institute for Cognitive Science Studies will collaboratively fund the project and lead subsequent dissemination and drug abuse and HIV risk reduction efforts in Iran.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Dependence

Exclusion Criteria:

* Dependence on alcohol, benzodiazepines or sedatives
* Suicide or homicide risk
* Psychotic disorder or major depression
* Inability to read or understand the protocol or assessment questions
* Life-threatening or unstable medical problems
* Greater than 3 times normal liver enzymes (AST, GGT)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Time to resumption of heroin use | 26 weeks
Time to relapse | 26 weeks
Maximum consecutive weeks of opiate abstinence | 26 weeks
Reduction of HIV risks | 26 weeks

SECONDARY OUTCOMES:
Addiction-related functional status | 26 weeks
Adverse events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Schottenfeld, M.D., Principal Investigator — Yale University; Azarakhsh Mokri, M.D., Study Director — Rouzbeh Hospital, Tehran, Iran
Locations (2):
- Yale University School of Medicine, New Haven, Connecticut, United States
- Institute for Cognitive Studies, Tehran, Iran